CLINICAL TRIAL: NCT02401594
Title: A Multicentre, Randomised, Double-blind, Controlled, Phase IIIb Study to Assess the Efficacy and Safety of Rivaroxaban 10mg od Versus Enoxaparin 4000 UI for VTE PROphylaxis in NOn Major Orthopaedic Surgery
Brief Title: PROphylaxis in NOn Major Orthopaedic Surgery
Acronym: PRONOMOS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Remaining outdated treatments and additional costs too high for new manufacturing
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1408143; 2015-000981-70 (EudraCT Number)
Record Dates: First submitted 2015-03-06; First posted 2015-03-30 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Non-major Orthopaedic Surgery
Keywords: Non-major orthopaedic surgery; deep vein thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Rivaroxaban treatment (Experimental): Rivaroxaban active substance plus a placebo of enoxaparin
  Interventions: Drug: Rivaroxaban
- Grouyp 2: Enoxaparine treatment (Active Comparator): Enoxaparin active substance plus a placebo tablet of Rivaroxaban
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban — 10 mg once daily of Rivaroxaban active substance (10 mg tablet) plus a placebo syringe of enoxaparin 4000 UI once daily
  Other Names: Group 1:
  Arms: Group 1: Rivaroxaban treatment
Drug: Enoxaparin — A syringe of enoxaparin active substance 4000 UI once daily plus a placebo tablet of Rivaroxaban 10 mg.
  Other Names: Group 2:
  Arms: Grouyp 2: Enoxaparine treatment

SUMMARY:
PRONOMOS is an international multicentre, interventional, parallel, randomised, double-blind non-inferiority study comparing rivaroxaban 10mg od to an active comparator, enoxaparin 4000 UI od in 4040 valid subjects requiring orthopaedic surgery (except low risk such material removal foot surgery or hallux valgus without patient risk factor [6], and major orthopaedic surgeries for femoral neck and trochanteric fractures, THR, TKR)

Pre-randomization treatment with LMWH anticoagulant is allowed for a maximum duration of 24 hours. However, only a single pre-randomization dose of LMWH is allowed. After randomization, patients allocated to the rivaroxaban arm will receive rivaroxaban 10 mg once-daily started 6-10 hours provided haemostasis has been established after surgery or 24h hours after LMWH injection if needed for the intended treatment duration of 2 to 12 weeks based on medical judgment (according to immobilization). Patients allocated to the comparator arm will receive enoxaparin once daily for the same intended treatment duration. All patients will have a 30-day observational period after cessation of treatment.

DETAILED DESCRIPTION:
Major orthopedic surgery (hip, knee replacements and hip fracture) represents only a small part of all orthopaedic surgery procedures. Procedures for trauma patients and orthopaedic lower limb surgery without trauma are much more frequent (tibia osteotomy, arthrodesis, ligament repair….).

The incidence of trauma patients requiring surgery and prolonged immobilisation is rising, mainly because of the increasing popularity of recreational sports. However, the epidemiology and prevention of VTE after such injuries have been poorly studied. The combination of limb surgery with or without trauma in orthopaedic surgery is responsible for an increase in venous thromboembolism (VTE). Usually, surgery of lower limb is considered as moderate or high risk for DVT with different duration related to immobilisation. For instance tibia osteotomy is at very high risk during at least 6 weeks and knee arthroscopy for ligament repair is at moderate risk during 10 days. However LMWH is recommended in both surgeries. Non-major orthopaedic surgery represents a major additional risk factor by itself; therefore such patients undergoing surgery deserve to receive VTE prophylaxis.

Rivaroxaban is a new oral anticoagulant developing a potent anti-Xa activity. In major orthopaedic surgery, it has shown to be more effective and as safe as LMWH (Enoxaparin 4000 IU once daily) in THR and TKR patients (RECORD program). Up to now, pending the limited number of surgical settings in which it has been developed in orthopaedic surgery, it is only approved for the prevention of venous thromboembolism (VTE) in THR and TKR procedures, which represent only 20% of all orthopaedic interventions. Non-major elective lower limb surgery and traumatology population is younger as compared to prosthetic orthopaedic surgery patients. Fewer VTE and cardiovascular events are to be feared. These patients receive quite often injectable thromboprophylaxis for a total duration lying between approximately 6 weeks to 3 months. In the one hand, the risk of major bleeding is low in this younger population. On the other hand, compliance and cost should be in favour of Rivaroxaban, because no injection and no platelets counts are needed.

The results of Xamos descriptive sub-analysis in non-elective (fracture related) orthopaedic surgery are consistent with the overall results of Xamos and are in favour of further investigations in this area. In this small subset of patients (n=790), the incidence of symptomatic thromboembolic events observed was low in patients treated with Xarelto and the overall frequency of treatment emergent major bleedings was low in both groups and serious adverse events occurred less frequently in patients treated with Xarelto. Therefore, collection of clinical data in this population is needed and awaited by many orthopaedic surgeons and anaesthetists in charge of VTE prophylaxis.

The population with femoral neck and trochanteric fracture is a specific one with different characteristics, elderly, frail and with a higher bleeding risk. This population will be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form,
2. Age ≥ 18 years,
3. Hospitalised for non-major orthopaedic surgery and requiring thromboprophylaxis according to the investigator's judgement on VTE risk such Achilles' repair, hip (except femoral neck and trochanteric fracture), knee, tibial plateau, femur (non femoral head), tibial and ankle fractures and tibial osteotomy, tibial transposition, arthrodesis of leg articulation, ligament repair of the knee or the ankle or any elective orthopaedic limb surgery requiring thromboprophylaxis).

Exclusion Criteria:

1. Major orthopaedic surgery Hip and Knee replacement, femoral neck and trochanteric fractures, spine surgery,
2. Low risk surgery without patient VTE risk: foot surgery (Hallux Valgus), material removal,
3. Delay between hospitalisation and randomisation greater than two days,
4. Women of childbearing potential not using a reliable contraceptive method throughout the study period (a list of reliable contraceptive methods is provided in the accompanying SPM),
5. Women pregnant or breast-feeding during the study period,
6. Body weight less than 50 kg (to avoid bleeding over risk) or over 120 kg,
7. Long term treatment with VKA therapy or NOAC,
8. Concomitant treatment with clopidogrel, prasugrel and ticagrelor,
9. Platelet count < 100 Giga/L,
10. Documented history of acquired or inherited bleeding disorder (e.g., von Willebrand's disease),
11. Severe renal failure with calculated creatinine clearance (Cockcroft Formula) < 30 mL/min,
12. Severe hepatic insufficiency with prothrombin time < 60% or liver impairment associated with coagulation disorders,
13. History of thrombocytopenia,
14. Any other current significant medical condition that might interfere with treatment evaluation according to the investigator's judgement,
15. Known hypersensitivity or other severe reaction to any component of the investigational medicinal product(s),
16. Participation in another clinical study involving an investigational medicinal product within 30 days prior to inclusion or concomitantly with this study,
17. Active bleeding or contraindication to anticoagulant therapy
18. Chronic alcoholic intoxication,
19. Anticipated poor compliance of subject with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3608 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Major VTE | From date of randomization until the date of the end of the treatment period (up to 3 months maximum).
  composite of proximal DVT (asymptomatic and symptomatic) assessed by ultrasonography, symptomatic events (distal and proximal DVT, PE) and VTE related deaths.
  The treatment period ranges from 15 days to 3 months depending on the type of surgery

SECONDARY OUTCOMES:
Major bleeding | From date of randomization until the date of the end of the treatment period (up to 3 months maximum).
  bleeding event that meets at least one of the following criteria [5]:
  * fatal bleeding;
  * critical bleeding (intracranial, intraocular, intraspinal, pericardial, retroperitoneal);
  * clinically overt bleeding (at surgical or extrasurgical site) associated with a decrease in the haemoglobin level of more than 2 g/dL (20 g/l; 1.24 mmol/L) compared with the pre-randomization level;
  * clinically overt bleeding (at surgical or extrasurgical site) leading to transfusion of two or more units of whole blood or packed cells;
  * bleeding located at the surgical site and leading to re-operation or to any unusual medical intervention or procedure for relief (e.g. draining or puncture of an haematoma at the surgical site, transfer to an ICU or emergency room) The treatment period ranges from 15 days to 3 months depending on the type of surgery
Clinically relevant non-major bleeding | From date of randomization until the date of the end of the treatment period (up to 3 months maximum)..
  overt bleeding not meeting the criteria for major bleeding and corresponds to any bleeding necessitating medical intervention or a specific, unscheduled consultation or treatment discontinuation, or resulting in a deterioration of the subject's quality of life. Some examples of clinically significant bleeding are given below:
  * Epistaxis that lasts more than five minutes or recurrent or necessitates packing,
  * Spontaneous macroscopic haematuria or haematuria lasting more than 24 hours after instrumentation,
  * Gastrointestinal haemorrhage (melena or rectorrhagia),
  * Haemoptysis,
  * Subcutaneous haematoma > 100 cm². The treatment period ranges from 15 days to 3 months depending on the type of surgery
Overt thrombocytopenia | From date of randomization until the date of the end of the treatment period (up to 3 months maximum)..
  platelet count <100 giga/L or fall ≥ 50% of the platelet count as compared with the first post-operative count which will be done as local lab for all centres The treatment period ranges from 15 days to 3 months depending on the type of surgery
Mortality | From date of randomization until the date of the end of the treatment period (up to 3 months maximum)..
  All cause mortality The treatment period ranges from 15 days to 3 months depending on the type of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAMAMA, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Nadia ROSENCHER, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Patrick MISMETTI, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (38):
- France (38):
  - CHU AMIENS Picardie, Amiens
  - CHU Angers, Angers
  - Clinique Générale d'ANNECY, Annecy
  - CHU BESANCON- Hôpital Jean Minjoz, Besançon
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Médipôle de Savoie, Challes-les-Eaux
  - Clinique Léonard de Vinci, Chambray-lès-Tours
  - CHU de Dijon- Bocage, Dijon
  - Hôpitaux Universitaires de Strasbourg C.C.O.M, Illkirch-Graffenstaden
  - CHU de Grenoble 6 Hôpital Michallon, La Tronche
  - Chu Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHRU Lille -Hôpital Roger Sallengro, Lille
  - CHU Dupuytren, Limoges
  - Ch Lyon Sud Pierre Benite, Lyon
  - Chu Marseille La Timone, Marseille
  - Ch Les Chanaux, Mâcon
  - CHU de MONTPELLIER - Lapeyronnie, Montpellier
  - CHRU NANTES - Hôtel Dieu, Nantes
  - CHU Carémeau, Nîmes
  - Clinique ARAGO, Paris
  - GH Paris Saint-Joseph, Paris
  - Hopital Cochin, Paris
  - Hopital Europeen Georges POMPIDOU, Paris
  - Ch Paris Pitie Salpetriere, Paris
  - Ch Saint Louis-Lariboisiere, Paris
  - CHU Bordeaux, Pessac
  - Polyclynique de Poitiers, Poitiers
  - CHU de Reims - Hôpital MAsion Blanche, Reims
  - Hôpital Robert Debré, Reims
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - CHU de SAINT-ETIENNE, Saint-Etienne
  - Clinique de la Mutualiste, Saint-Etienne
  - Chp Saint Gregoire, Saint-Grégoire
  - Polyclinique Du Parc, Saint-Saulve
  - CHRU de Strasbourg- Hôpital Hautepierre, Strasbourg
  - Clinique Médipôle, Toulouse
  - CHU Toulouse - Hôpital Pierre-Paul Riquet, Toulouse

REFERENCES:
- [Derived] Samama CM, Laporte S, Rosencher N, Girard P, Llau J, Mouret P, Fisher W, Martinez-Martin J, Duverger D, Deygas B, Presles E, Cucherat M, Mismetti P; PRONOMOS Investigators. Rivaroxaban or Enoxaparin in Nonmajor Orthopedic Surgery. N Engl J Med. 2020 May 14;382(20):1916-1925. doi: 10.1056/NEJMoa1913808. Epub 2020 Mar 29. PMID 32223113